CLINICAL TRIAL: NCT03492879
Title: Non Invasive Electrical Impedance Technology (EIT) for Diagnosing Liver Diseases Severity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Ziv Ben-Ari MD (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Ziv Ben-Ari MD, Head of liver diseases center, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-17-4351-CTIL
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Chronic Liver Disease; Fibrosis, Liver; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biopsy: Routine tests & EIT Technology (Experimental): The patients will undergo a routine liver biopsy and also routine liver Ultrasonography, Shear wave elastography and Electrical Impedance Technology (EIT).
  Interventions: Device: EIT Technology
- Routine tests & EIT Technology (Experimental): The patients will undergo a routine liver Ultrasonography, Shear wave elastography and Electrical Impedance Technology (EIT).
  Interventions: Device: EIT Technology
- NASH : Routine tests & EIT Technology (Experimental): The patients will undergo a routine liver Ultrasonography, Shear wave elastography and quantification of liver steatosis using the Electrical Impedance Technology (EIT).
  Interventions: Device: EIT Technology

INTERVENTIONS:
Device: EIT Technology — Electrical Impedance Technology is a non-invasive imaging method who is being tested for evaluation of liver fibrosis stage

SUMMARY:
The aims of this study are to assess the performance of the non-invasive Electrical Impedance Technology (EIT) in evaluating the liver fibrosis stage in patients with chronic liver diseases, in comparisons with a liver biopsy and/or Shear wave elastography and Liver Ultrasonography.

The second aim is comparing between Liver Ultrasonography and Electrical Impedance Technology (EIT) to quantify the hepatic steatosis grade in patients with Non Alcoholic Fatty Liver Disease (NAFLD) .

DETAILED DESCRIPTION:
The study will include 210 patients with chronic liver diseases. Relevant clinical data such as sex, age, weight, height, alcohol intake, medical history and routine lab results will be collected.

The study will include three groups:

1. Patients with indication for liver biopsy will undergo a routine liver biopsy and also routine liver Ultrasonography, Shear wave elastography and Electrical Impedance Technology (EIT) (70 patients).
2. Patients with chronic liver diseases will undergo routine liver Ultrasonography, Shear wave elastography and Electrical Impedance Technology (EIT) (70 patients).
3. Patients with Non Alcoholic Fatty Liver Disease will undergo routine liver Ultrasonography, Shear wave elastography and quantification of liver steatosis using the Electrical Impedance Technology (EIT) (70 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver diseases

Exclusion Criteria:

* Patients who don't have chronic liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the liver fibrosis stage using Electrical Impedance Technology (EIT) | Each technology will be performed once in 1 year
  Comparing EIT fibrosis stage result to fibrosis stage result of validated thechnologies

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Ben-Ari, MD, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: Undecided